CLINICAL TRIAL: NCT00028665
Title: Randomized Phase II Trial of B-Lymphocyte Purging of Autologous Peripheral Blood Progenitor Cells in Patients With B-Cell Non-Hodgkin's Lymphoma
Brief Title: Cyclophosphamide W/or W/Out Rituximab and Peripheral Stem Cell Transplantation in Patients With Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Omer Koc, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1499; P30CA043703 (NIH); CWRU1499 (Other: Case Comprehensive Cancer Center); CWRU-030040; NCI-G01-2040
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Rituximab; Carmustine; Cisplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: with rituximab IV (Experimental)
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: carmustine; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- Arm II: without rituximab IV (Active Comparator)
  Interventions: Biological: filgrastim; Drug: carmustine; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Beginning 36-48 hours after the completion of cyclophosphamide, patients receive filgrastim (G-CSF) subcutaneously (SC) daily until blood counts recover. Patients receive G-CSF SC daily beginning 4 hours after completion of PBSC infusion and continuing until neutrophil engraftment.
Biological: rituximab — rituximab IV over 2-5 hours on days 1, 8, and 15
  Arms: Arm I: with rituximab IV
Drug: carmustine — After completion of PBSC collection, patients receive high-dose chemotherapy comprising carmustine IV on days -7 to -3
Drug: cisplatin — After completion of PBSC collection, cisplatin IV for 3 days during days -7 to -3.
Drug: cyclophosphamide — cyclophosphamide IV over 3-6 hours on day 16.
Drug: etoposide — After completion of PBSC collection, etoposide IV for 3 days during days -7 to -3.
Procedure: bone marrow ablation with stem cell support — Patients then undergo peripheral blood stem cell (PBSC) collection.
Procedure: peripheral blood stem cell transplantation — Arm I: Patients receive unmanipulated PBSCs on day 0. Arm II: Patients receive CD34 cell-enriched PBSC on day 0.
Radiation: radiation therapy — Patients may undergo involved-field radiotherapy to active or previously bulky (more than 5 cm) tumors daily for 7-10 days.

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known if combining rituximab with cyclophosphamide is more effective than cyclophosphamide alone in stimulating peripheral stem cells for transplantation.

PURPOSE: This randomized phase II trial is studying how well giving cyclophosphamide with or without rituximab followed by chemotherapy and peripheral stem cell transplantation works in treating patients with recurrent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of mobilization therapy with or without rituximab on hematopoietic stem cells, B and T lymphocytes, and natural killer cells in patients with advanced or recurrent B-cell non-Hodgkin's lymphoma.
* Compare the effects of B-lymphocyte purging using concurrent rituximab and mobilization therapy vs a CD34+ cell enrichment device on hematopoietic stem cells, B and T lymphocytes, and natural killer cells in the peripheral blood stem cell (PBSC) infusates.
* Compare the effect of these purging regimens on tumor cell content of PBSC infusates.
* Compare the effects of these regimens on myeloid and lymphoid engraftment after high-dose chemotherapy and autologous PBSC infusion in these patients.
* Compare post-transplantation infection complications in patients treated with these regimens.
* Compare the response and relapse-free survival of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive mobilization therapy comprising rituximab IV over 2-5 hours on days 1, 8, and 15 and cyclophosphamide IV over 3-6 hours on day 16. Beginning 36-48 hours after the completion of cyclophosphamide, patients receive filgrastim (G-CSF) subcutaneously (SC) daily until blood counts recover. Patients then undergo peripheral blood stem cell (PBSC) collection.

After completion of PBSC collection, patients receive high-dose chemotherapy comprising carmustine IV on days -7 to -3 and etoposide IV and cisplatin IV for 3 days during days -7 to -3. Patients may undergo involved-field radiotherapy to active or previously bulky (more than 5 cm) tumors daily for 7-10 days.

Patients receive unmanipulated PBSCs on day 0. Patients receive G-CSF SC daily beginning 4 hours after completion of PBSC infusion and continuing until neutrophil engraftment.

* Arm II: Patients receive mobilization therapy comprising cyclophosphamide and G-CSF and high-dose chemotherapy comprising carmustine, etoposide, and cisplatin as in arm I. Patients may also undergo involved-field radiotherapy as in arm I. Patients receive CD34 cell-enriched PBSC on day 0 followed by G-CSF as in arm I.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell non-Hodgkin's lymphoma (NHL)

  * Indolent or aggressive histology
  * No small lymphocytic lymphoma, Burkitt's lymphoma, or small lymphocytic non-Burkitt's lymphoma
* CD20-positive and/or CD19-positive by immunohistochemistry or flow cytometry
* Second or greater remission allowed

  * Partial remission, relapse, or refractory disease must have measurable tumor
* Eligible for high-dose therapy followed by autologous peripheral blood stem cell transplantation
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age:

* 12 to 65

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,200/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine clearance at least 60 mL/min
* No renal dysfunction

Cardiovascular:

* LVEF at least 40%
* No cardiac dysfunction
* No myocardial infarction within the past 3 months

Pulmonary:

* FEV_1 greater than 60%
* DLCO at least 60% of predicted
* No pulmonary dysfunction
* No asthma

Other:

* HIV negative
* No significant organ dysfunction
* No severe comorbid condition
* No uncontrolled diabetes
* No severe or active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* No prior immunotherapy

Chemotherapy:

* No prior high-dose chemotherapy with or without peripheral blood stem cell transplantation
* No more than 3 prior chemotherapy regimens for NHL
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Not specified

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-06; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Total CD34 cells | measured at baseline, at time of harvests, days 42 and 90 after the transplant, and 6 and 12 months after the transplant
T and B lymphocyte counts | measured at baseline, at time of harvests, days 42 and 90 after the transplant, and 6 and 12 months after the transplant
Disease response | measured at 4 weeks after the transplant
Engraftment | measured at days 42 and 90 after the transplant, and 6 and 12 months after the transplant

CONTACTS AND LOCATIONS:
Overall Officials: Omer N. Koc, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio, United States